CLINICAL TRIAL: NCT06648382
Title: Pilot Test of a Self-Directed Psychotherapy Program for Premenstrual Disorders
Brief Title: Pilot Study of the 'Thriving With PMDs' Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: International Association for Premenstrual Disorders (Unknown)
Responsible Party: Principal Investigator, Jennifer Gordon, Associate professor, University of Regina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB 2024-916; 6541 (Other Grant/Funding Number: Saskatchewan Health Research Foundation)
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-10

CONDITIONS: Premenstrual Disorder; Premenstrual Dysphoric Disorder
Keywords: Psychotherapy; Premenstrual disorder; Premenstrual dysphoric disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Self-directed psychotherapy program (Experimental): The intervention consists of receiving 11 videos that are 10-15 minutes in length along with a workbook containing homework exercises. Participants are instructed to watch the videos over the course of two menstrual cycles: the first 6 during the first cycle and the last 5 during the second cycle. Each module focuses on a different skill inspired by cognitive behavioral therapy and dialectical behavior therapy.
  Interventions: Behavioral: Self-directed psychotherapy program for premenstrual disorders

INTERVENTIONS:
Behavioral: Self-directed psychotherapy program for premenstrual disorders — The intervention consists of receiving 11 videos that are 10-15 minutes in length along with a workbook containing homework exercises. Participants are instructed to watch the videos over the course of two menstrual cycles: the first 6 during the first cycle and the last 5 during the second cycle. Each module focuses on a different skill inspired by cognitive behavioral therapy and dialectical behavior therapy.

SUMMARY:
This study is testing a self-help mental health program that was designed to help people cope with the challenges of living with a premenstrual disorder. Individuals with a premenstrual disorder - either premenstrual dysphoric disorder or premenstrual exacerbation of depression - will track their daily symptoms for two menstrual cycles before they complete the program, throughout the two-cycle program, and for an additional two cycles after accessing the program. This will allow the research team to compare their symptoms before and after accessing the program.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-42
* Either meeting diagnostic criteria for premenstrual dysphoric disorder (to be confirmed by researchers through daily symptom ratings for two menstrual cycles) or major depressive disorder with perimenstrual exacerbation (i.e. at least a 30% increase in 4 symptoms in the perimenstrual phase)

Exclusion Criteria:

* Taking oral contraceptives
* Currently in psychotherapy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pre-to-post changes in perimenstrual Daily Record of Severity of Problems (DRSP) score (range of scores = 24-144) | Baseline, 1 month post-intervention, 2 months post-intervention
  Perimenstrual DRSP score during the two post-intervention menstrual cycles relative to the two pre-intervention menstrual cycles

CONTACTS AND LOCATIONS:
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
The data collected is sensitive in nature - there are many questions about suicidality and urges to self harm as well as experiences with traumatic events. We do not want to make participants feel uncomfortable by making their data publically available.